CLINICAL TRIAL: NCT05621720
Title: Adopting a Health-social Partnership Program to Promote Health and Self-care Management Among Older Adults in the Community: an Effectiveness-implementation Hybrid Design
Brief Title: Adopting a Health-social Partnership Program to Promote Health and Self-care Management Among Older Adults in the Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Frances Kam Yuet WONG, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20210401002
Record Dates: First submitted 2022-06-13; First posted 2022-11-18 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Healthy Aging
Keywords: Community-dwelling older adults; Self-care; Health and social partnership
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the outcome(s) of interest would be blinded from having knowledge of the intervention and control group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in the intervention group will receive a 3-moth community-based health-social partnership program (C-HSPP) led by a nurse case manager, and supported by social workers and community workers.
  Interventions: Other: Case management
- Control group (Other): Subjects in the control group will receive usual community services and a monthly social control call from trained community workers.
  Interventions: Other: Social control call and usual are

INTERVENTIONS:
Other: Case management — On enrolment, the nurse case manager will perform the initial comprehensive assessment based on the Omaha domains of environment, psychosocial, physiological and health-related behavior. The nurse case manager will execute the intervention scheme of teaching, guidance & counseling, treatments & procedure, case management, and/or surveillance, with the mutual goal set with clients to promote health and self-efficacy. Home visits and telephone calls will be employed. The referral network to health and social service will be activated as appropriate.
  Arms: Intervention group
Other: Social control call and usual are — Subjects in the control group will receive usual community service. in addition, a monthly social control call from trained community workers will be given to rule out the possible social effects of the intervention. These social calls will not be related the participants' health condition nor delivery of any health information.
  Arms: Control group

SUMMARY:
Hong Kong has notably the longest life expectancy in the world. Ever-increasing demand and challenges are posing to the healthcare, social welfare, and elderly care service system. As a global public health strategy to address the increasing burdens, there is a strong urge for an effective approach to enhance the health and self-care ability among the older adults dwelling in the community. Literature suggested that the effectiveness of community-based self-care management programs is inconclusive. In addition, though the concept of the health-social partnership has been widely promoted to improve primary care, literature addressed that the multiple barriers existed throughout the collaboration. More evidence should be sought in the local context to evaluate the effectiveness of self-care complex interventions program among older adults.

DETAILED DESCRIPTION:
This randomized type 2 effectiveness-implementation hybrid trial study aims to examine the effectiveness of a community-based health-social partnership program in promoting health and self-care management among older adults dwelling in the community and to explore the reach, adoption, implementation, maintenance aspects of the implementation process of the program in a real-life setting.

This study has two parts. The first part involves a cluster randomized controlled trial with a two-arm, matched-pairs, equivalent allocation ratio, and parallel design to examine the effectiveness of this study. Based on socio-economic status, community centers will be matched into three comparable pair sets, and further randomized into three intervention and control groups. A total of 788 subjects (394 in each arm) aged 60 or above, dwelling in the community, and cognitively competent will be recruited. Three-time interval outcome measures will be collected. The second part of this study is an implementation research design concerning the implementation process of the program in a real-life setting. Focus group interviews with different stakeholders will be conducted and meeting minutes, and archives of documents will be studied. Summative data will be analyzed in the RE-AIM framework.

The findings of this study are anticipated to shed some light on the effectiveness and implementation of integrated health-social service in Hong Kong context. It will make important contributions, not only to the individuals, but also to the policymakers and service providers advocating the concept of ageing in place and health-social partnership approach care. The informed the health-social partnership collaboration practice in real-world setting can facilitate the translation of research evidence into practice to tackle the health burdens and challenges.

ELIGIBILITY:
Inclusion Criteria:

* (i) People aged 60 or above
* (ii) Living within the service areas of respective community centers
* (iii) Cognitively competent with Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) with score ≥22

Exclusion Criteria:

* (i) Not communicable
* (ii) Not reachable by phone
* (iii) Not living at home
* (iv) Bed bound
* (v) With serious mental illness requiring hospitalization in recent 6 months
* (vi) Already engaged in similar structured health or social programs
* (vii) Will not stay in Hong Kong for the current three months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 788 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Self-efficacy | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  The General Self-Efficacy Scale (GSE), developed based on social cognitive theory, initially consisted of 20 items and was later refined to a 10-item version that has been translated into Chinese. The scale items are rated on a 4-point Likert scale, ranging from 1 (not at all true) to 4 (exactly true). The total score ranges from 10 to 40, with higher scores indicating greater self-efficacy, meaning a stronger belief in one's ability to handle various situations effectively.
Change in Instrumental Activities of Daily Living (IADL) | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  The instrumental activities of daily living is measured by Lawton Instrumental Activities of Daily Living (IADL) Scale-Chinese version, a four-point scale with 9-items of activities which include use of telephone, transportation, shopping, meal preparation, housework, handyman work, laundry, medication management, and money management. Each item rate trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the night responses. Higher score means a worse IADL.

SECONDARY OUTCOMES:
Change in quality of life | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Quality of Life will be assessed using the 12-item Short Form Health Survey, version 2, Chinese (HK) version (SF-12v2). This survey includes subscales for physical functioning, role limitations due to physical and emotional problems, mental health, bodily pain, general health, vitality, and social functioning. Scores are weighted according to standard scoring algorithms and benchmarked against general population norms, yielding two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), each on a scale from 0 to 100. Higher scores indicate better quality of life, with higher PCS and MCS scores reflecting better physical and mental health, respectively.
Change in self-report of pain | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Using numeric (0-10) pain rating scale to assess the pain level. 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Change in depression | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Using the 15-item Chinese version of the Geriatric Depression Scale (GDS) to assess depression level. The maximum score is 15 (higher score, more severe) with a cut-off point of 8 with high sensitivity and specificity for detection of depression
Change in activity of daily living | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Use of Modified Barthel Index-Chinese version to measure 10 basic activities of daily living function (feeding, dressing, grooming, bathing, toileting, bed-chair transfer, bladder and bowel control, ambulation and stair climbing).It is measured using a 5-point Likert scale from 1= totally dependent to 5= fully independent. Higher score means better in performing activity of daily living.
Change in health service utilization | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Measuring the number of attendance to government out-patient clinics (GOPC), and number of unscheduled visits to the emergency department and hospital admission.
Change in blood pressure | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Blood pressure measurement will be performed after 10 minutes of sitting rest. A standard electronic sphygmomanometer will be used to measure supine blood pressure on the right arm of each candidate (unless contraindicated). Both systolic and diastolic blood pressure will be measured. Individuals with an average BP 135/85mmHg based on readings in the morning and evening based on 6 consecutive days are considered to be hypertensive based on the Hong Kong Reference Framework for Hypertension Care for Adults in Primary Care Settings.
Change in body mass index | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  BMI will be measured by the calculation of weight/(height*height) based on a regularly calibrated weight scale and stadiometer when the subjects wear light clothing without shoes. Normal readings are within 18.5-23.
Change in fall incidence | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Asking the fall incidence in the past three months. A fall diary is suggested to completed.
Change in medication adherence | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Using 12-item Adherence to Refills and Medications Scale to the respondent's ability to take and refill all prescribed medications under different circumstances.The options vary from "none of the time" to "all of the time", with total scores ranging from 12-48 . Higher score means worse in adherence to refills and medication.
Change in capillary blood glucose | Baseline pre-intervention (T1), at three-month when the interventions are completed (T2), and three-month post-intervention (T3)
  Capillary blood glucose level will be measured by a standard capillary glucose meter.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Kam-Yuet Wong, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwok WYY, Wong FKY, Wong AKC, Bayuo J. Community-Based Health-Social Partnership Programme (C-HSPP) for enhancing self-care management among older adults: protocol for a hybrid effectiveness-implementation trial. BMC Public Health. 2025 May 7;25(1):1678. doi: 10.1186/s12889-025-22846-6. PMID 40335958